CLINICAL TRIAL: NCT06572072
Title: Effects of Negative Pressure Ventilation on Right Ventricular Function in Cardiological Patients With Reduced Right Ventricular Function.
Brief Title: Effects of Negative Pressure Ventilation on Right Ventricular Function in Cardiological Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Karlsburg Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Matthias Heringlake, Principal Investigator, Karlsburg Hospital
Other Study IDs: KAIKB-2024_1
Record Dates: First submitted 2024-08-07; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Negative Pressure Ventilation; Right Ventricular Dysfunction; Right Ventricular Failure
MeSH Terms: conditions — Ventricular Dysfunction, Right; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Negative Pressure Ventilation — Substitution of positive pressure ventilation by negative pressure ventilation

SUMMARY:
Patients receives induction of general anesthesia for interventional tricuspidal clipping and standard monitoring for this procedure including arterial and central venous line and transesophageal ultrasound. A cuirass for extrathoracal negative pressure ventilation is placed onto the chest but not switched on. During usual positive pressure ventilation a ventilatory, a hemodynamic and a 3D full volume ultrasounddataset of the right and left ventricle is recorded and severity of tricuspidal regurgitation examined. Afterwards negative pressure ventilation is started and positive pressure ventilation reduced as far as possible without reduction of tidal volumes. The same dataset of ventilation, hemodynamics and ultrasound is collected again during negative pressure ventilation. Afterwards the cuirass gets removed, study finished and everything proceeds as during standard procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients planned for tricuspidal clipping

Exclusion Criteria:

* ventilatory of hemodynamic instability
* fitting of cuirass not possible
* unavailability of examiner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients for tricuspidal clipping without an exclusion criterium
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
stroke volume index | 1 minute
  transesophageal ultrasound measurement

SECONDARY OUTCOMES:
RVEF | 1 minute
  transesophageal ultrasound measurement
LVEF | 1 minute
  transesophageal ultrasound measurement
volumes of chambers | 1 minute
  transesophageal ultrasound measurement
strain | 1 minute
  transesophageal ultrasound measurement
VC | 1 minute
  transesophageal ultrasound measurement
PISA | 1 minute
  transesophageal ultrasound measurement
EROA | 1 minute
  transesophageal ultrasound measurement
area of regurgitation of tricuspid valve | 1 minute
  transesophageal ultrasound measurement
arterial blood pressures | 1 minute
  hemodynamic measurements
venous blood pressures | 1 minute
  hemodynamic measurements
pulmonal blood pressures | 1 minute
  hemodynamic measurements
heart frequency | 1 minute
  hemodynamic measurements
tidal volume | 1 minute
  ventilatory measurements
minute volume | 1 minute
  ventilatory measurements
breathing rate | 1 minute
  ventilatory measurements
etCO2 | 1 minute
  ventilatory measurements
pO2 in the blood | 1 minute
  blood gases
pCO2 in the blood | 1 minute
  blood gases
Laktat | 1 minute
  blood gases
cerebral oximetry | 1 minute
  NIRS

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Karlsburg, Klinik für Anästhesiologie, Karlsburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No